CLINICAL TRIAL: NCT01684033
Title: Evaluation of the Effectiveness of Two Marketed Multi-Purpose Solutions for Silicone Hydrogel Contact Lenses - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: M-12-038; 1941/ALC
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Myopia; Hyperopia; Contact Lens Comfort
Keywords: multi-purpose solution; silicone hydrogel; contact lenses; comfort; Opti-Free; Biotrue
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PureMoist - Biotrue (Other): Opti-Free® PureMoist® MPDS used first, followed by Biotrue™ MPS. Each product used as indicated for 30 days with participant's habitual contact lenses.
  Interventions: Device: Opti-Free® PureMoist® MPDS; Device: Biotrue™ MPS; Device: Habitual contact lenses
- Biotrue - PureMoist (Other): Biotrue™ MPS used first, followed by Opti-Free® PureMoist® MPDS. Each product used as indicated for 30 days with participant's habitual contact lenses.
  Interventions: Device: Opti-Free® PureMoist® MPDS; Device: Biotrue™ MPS; Device: Habitual contact lenses

INTERVENTIONS:
Device: Opti-Free® PureMoist® MPDS
  Other Names: OPTI-FREE® PureMoist™
Device: Biotrue™ MPS
  Other Names: Biotrue™
Device: Habitual contact lenses — Silicone hydrogel contact lenses per participant's habitual brand, prescription, and replacement schedule worn on a daily wear basis for at least 8 hours a day, 5 days a week for the duration of the study. During the washout period, the contact lenses were worn on a daily disposable basis.

SUMMARY:
The purpose of this study was to evaluate the performance of Opti-Free® PureMoist® Multi-Purpose Disinfecting Solution (MPDS) compared to Biotrue™ Multipurpose Solution (MPS) in silicone hydrogel contact lens wearers.

DETAILED DESCRIPTION:
In this 2-period crossover study, eligible participants were randomized to either Opti-Free® PureMoist® Multi-Purpose Disinfecting Solution or Biotrue™ Multipurpose Solution in Period 1 for use with their habitual contact lenses, after which they switched to the alternate solution in Period 2. Each period was 30 days in length. A 2-day washout period during which participants refrained from using a multi-purpose contact lens solution preceded Period 1 and Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Wear single vision sphere silicone hydrogel contact lenses (CooperVision™ Biofinity®, Alcon® Air Optix® Aqua, Bausch+Lomb® PureVision™ or ACUVUE® Oasys™) on a daily wear basis (a minimum of 8 hours per day, 5 days a week) for at least one month prior to Visit 1;
* Willing to wear lenses on a daily wear basis (a minimum of 8 hours per day, 5 days a week) for the duration of the study, and wear lenses for 16 hours on two days during the study;
* Must have habitually used a Biguanide preserved multi-purpose solution (other than Biotrue) for at least 30 days prior to Visit 1;
* Vision correctable to 20/30 Snellen (feet) or better in each eye at distance with pre-study contact lenses at Visit 1;
* Have access, capability and willingness to review and answer text messages;
* Read, sign, and date IRB/IEC approved informed consent and privacy document before enrollment;
* Willing to follow the study procedures and visit schedule;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Need to wear lenses on an extended wear (i.e. overnight) basis during the study;
* Known sensitivity or intolerance to Biguanide, polyquaternium-1 (POLYQUAD), or ALDOX preserved lens care products;
* Monocular (only one eye with functional vision) or fit with only one lens;
* Wearing toric or multifocal contact lenses or fit with monovision;
* Use of additional lens care products other than a Biguanide preserved multipurpose solution such as daily or enzyme cleaners within the one week prior to Visit 1;
* Use of topical ocular over-the-counter (OTC) or prescribed topical ocular medications, with the exception of rewetting drops, within 7 days prior to Visit 1;
* Abnormal ocular condition observed during the Visit 1 slit-lamp examination;
* Current or history of ocular infections or severe inflammation within 6 months prior to Visit 1;
* Ocular surgery within the 12 months prior to Visit 1;
* Participation in any other clinical trial within 30 days of enrollment;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Lemp, MS, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 study centers located in the US, 3 study centers located in the UK, and 2 study centers located in Germany.
Pre-assignment Details: Of the 207 enrolled, 9 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants who were exposed to a study regimen (test or control) (198).
Groups:
- PureMoist - Biotrue: Opti-Free® PureMoist® MPDS, followed by Biotrue™ MPS. Each product used as indicated for 30 days with participant's habitual contact lenses.
- Biotrue - PureMoist: Biotrue™ MPS, followed by Opti-Free® PureMoist® MPDS. Each product used as indicated for 30 days with participant's habitual contact lenses.
Period: Period 1, First 30 Days
Arm/Group | PureMoist - Biotrue | Biotrue - PureMoist
Started | 99 | 99
Completed | 95 | 98
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Noncompliance | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Period 2, Second 30 Days
Arm/Group | PureMoist - Biotrue | Biotrue - PureMoist
Started | 95 | 98
Completed | 94 | 98
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who were exposed to a study regimen (test or control).
Groups:
- PureMoist / Biotrue: Opti-Free® PureMoist® MPDS and Biotrue™ MPS used during Period 1 and Period 2 in randomized order in crossover assignment.
Arm/Group | PureMoist / Biotrue
Number analyzed (Participants) | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining
Description: Corneal staining in both eyes was assessed during slit lamp examination using flourescein dye. Each of five corneal regions (central, nasal, temporal, inferior, and superior) was graded on a scale from 0 (none) to 4 (patch). The corneal fluorescein staining score was calculated as the total of the five regions. The score ranged from 0 (no staining in any region) to 20 (patch staining in all five regions). The corneal staining of the worse eye was analyzed.
Time Frame: Day 30
Population: This analysis population group includes all participants who were exposed to both treatment regimens.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PureMoist: Opti-Free® PureMoist® MPDS used during Period 1 or Period 2 for 30 days with participant's habitual contact lenses.
- Biotrue: Biotrue™ MPS used during Period 1 or Period 2 for 30 days with participant's habitual contact lenses.
Arm/Group | PureMoist | Biotrue
Number analyzed (Participants) | 192 | 192
Units on a scale | 1.9 (2.30) | 2.8 (2.62)

2. Primary Outcome: Change From Baseline in Corneal Staining at Day 30
Description: as for outcome 1
Time Frame: Baseline (Day 0), Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PureMoist | Biotrue
Number analyzed (Participants) | 192 | 192
units on a scale | 0.7 (2.59) | 1.6 (2.91)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected for the duration of the study (4 months). AEs were elicited by non-direct questioning of the participant and spontaneous reporting by the participant. AEs were recorded at every visit.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device. This analysis population includes all participants who were exposed to a study regimen (test or control), based on treatment-specific exposure.
Arm/Group | PureMoist | Biotrue
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/194
Other Adverse Events (participants affected / at risk) | 0/196 | 0/194

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.